CLINICAL TRIAL: NCT00393510
Title: An Evidence Base Study on the Clinical Effects of Integrated Western Medicine and Traditional Chinese Medicine for Diabetic Foot Ulcer Treatment
Brief Title: Herbal Preparation Used as Adjuvant Therapy on Diabetic Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: The Institute of Chinese Medicine, CUHK, The Institute of Chinese Medicine, CUHK
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRE-8342
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Results first posted 2010-07-01 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Diabetic Foot Ulcer; Amputation
Keywords: Diabetic Foot Ulcer; Traditional Chinese Medicine
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Chinese Medicine (Active Comparator): 12 herbals formulation was given as an adjuvant therapy for the patients orally twice a day.
  Interventions: Drug: TCM
- Placebo (Placebo Comparator): Placebo was made with starch and colouring materials. Given to patient orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TCM — The Decoction is taken orally, twice a day, treatment period is 24 weeks The herbal formulation or a placebo was given as an adjuvant therapy for the treatment of the unhealing ulcers in these diabetic patients.
  The formula consisted of 12 herbs, viz:
  Radix astragali, Rhizoma atractylodis marcocephalae, Radix stephaniae tetrandrae, Radix polygoni multiflori, Radix rehmanniae, Radix smilax china, Fructus corni, Rhizoma dioscoreae, Cortex moutan, Rhizoma alismatis, Rhizoma smilacis glabrae, and Fructus schisandrae
  Arms: Traditional Chinese Medicine
Drug: Placebo — Placebo taking orally, twice a day, 24 week treatment period The herbal formulation or a placebo was given as an adjuvant therapy for the treatment of the unhealing ulcers in these diabetic patients.
  The placebo was made with starch and colouring materials.
  Arms: Placebo

SUMMARY:
Chronic foot ulcers occurring among diabetic patients are difficult to heal. The frequent elderly age with co-morbidities, vascular insufficiencies, peripheral neuropathies and super imposed infections, all contribute towards the chronicity and failure of treatment. Preserving the ulcerated limb is the patients' wish. On the other hand, an infected ulcer that never heals just unnecessarily prolongs suffering. Nevertheless, patients earnestly like to try all methods of healing before accepting amputation.

Objective:To determine whether a course of herbal preparation used as an adjuvant therapy for diabetic patients suffering from chronic foot ulcers may promote healing so that major leg amputation can be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Well Controlled diabetic state
* Presence of gangrene or non-healing ulcer in diabetic patients over the foot or feet. Infection should be well controlled.
* Good glycaemic control

Exclusion Criteria:

* Pregnant women and women at risk of conception
* Patients taking digitalis glycosides
* Patients with abnormal liver function tests
* Patients with plasma creatinine great then 150 umol/l or unstable renal function
* Poorly controlled Diabetes Mellitus
* Uncontrolled infection
* History of adverse reaction to herbal medicine
* Unstable medical conditions
* Non-compliance with regime

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2000-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leung Ping Chung, MD, Principal Investigator — Dept. of Orthopaedics & Traumatology, CUHK
Locations (2):
- China (2):
  - Department of Orthopaedics & Traumatology, Prince of Wales hospital, Hong Kong
  - Department of Orthopaedics and Traumatology, Kwong Wah Hospital, Hong Kong

REFERENCES:
- [Background] Levin ME. Diabetic foot ulcers: pathogenesis and management. J ET Nurs. 1993 Sep-Oct;20(5):191-8. PMID 8110884
- [Background] Nelzen O, Bergqvist D, Lindhagen A. High prevalence of diabetes in chronic leg ulcer patients: a cross-sectional population study. Diabet Med. 1993 May;10(4):345-50. doi: 10.1111/j.1464-5491.1993.tb00077.x. PMID 8508618
- [Background] Steed DL, Goslen JB, Holloway GA, Malone JM, Bunt TJ, Webster MW. Randomized prospective double-blind trial in healing chronic diabetic foot ulcers. CT-102 activated platelet supernatant, topical versus placebo. Diabetes Care. 1992 Nov;15(11):1598-604. doi: 10.2337/diacare.15.11.1598. PMID 1468291
- [Background] Ahlgren SC, Levine JD. Protein kinase C inhibitors decrease hyperalgesia and C-fiber hyperexcitability in the streptozotocin-diabetic rat. J Neurophysiol. 1994 Aug;72(2):684-92. doi: 10.1152/jn.1994.72.2.684. PMID 7983528
- [Background] Bazan NG, Gordon WC, Marcheselli VL, Lukiw WJ, Duhault J, Koenig-Berard E, Linn DM, DeCoster MA, Mukherjee PK. Experimental models and their use in studies of diabetic retinal microangiopathy. Therapie. 1997 Sep-Oct;52(5):447-51. PMID 9501573
- [Background] Diemel LT, Brewster WJ, Fernyhough P, Tomlinson DR. Expression of neuropeptides in experimental diabetes; effects of treatment with nerve growth factor or brain-derived neurotrophic factor. Brain Res Mol Brain Res. 1994 Jan;21(1-2):171-5. doi: 10.1016/0169-328x(94)90391-3. PMID 7513041
- [Background] Follansbee MH, Beyer KH Jr, Griffith JW, Vesell ES. Studies on pyrazinoylguanidine. 5. Temporal effects over 24 weeks demonstrating attenuation of diabetic nephropathy in STZ-diabetic rats. Pharmacology. 1997 May;54(5):241-55. doi: 10.1159/000139492. PMID 9380770
- [Background] Kunjathoor VV, Wilson DL, LeBoeuf RC. Increased atherosclerosis in streptozotocin-induced diabetic mice. J Clin Invest. 1996 Apr 1;97(7):1767-73. doi: 10.1172/JCI118604. PMID 8601643
- [Background] Liu S, Barac-Nieto M. Renal protein degradation in streptozotocin diabetic mice. Diabetes Res Clin Pract. 1997 Jan;34(3):143-8. doi: 10.1016/s0168-8227(96)01353-8. PMID 9069565
- [Background] Mavrikakis ME, Sfikakis PP, Kontoyannis D, Horti M, Kittas C, Koutras DA, Raptis SA. Macrovascular disease of coronaries and cerebral arteries in streptozotocin-induced diabetic rats. A controlled, comparative study. Exp Clin Endocrinol Diabetes. 1998;106(1):35-40. doi: 10.1055/s-0029-1211947. PMID 9516057
- [Background] Zochodne DW, Murray MM, van der Sloot P, Riopelle RJ. Distal tibial mononeuropathy in diabetic and nondiabetic rats reared on wire cages: an experimental entrapment neuropathy. Brain Res. 1995 Nov 6;698(1-2):130-6. doi: 10.1016/0006-8993(95)00876-r. PMID 8581471
- [Background] Wagner EW. Classification of neuropathic foot problems AAOS instructional lecture 28 St. Louis Mosby 1979 p143-165
- [Background] Brodsky JW. Diabetic Foot Surgery of Foot and Ankle. St. louis Mosby 1992, p1361-1467
- [Background] Conn, H.M., M.A. and Emmel, V.M. Staining Procedures. Williams and Wilkins Co., Baltimore, 289 pp.m (1960)
- [Background] Professor P.C. Leung. Limb Salvage for Diabetic ulceration with Traditional Chinese Techniques. Pacific, BioTech News. Vol.1 No.31 1998, Singapore
- [Background] J.Y.Shi, Collected publications on the applicatioin of Shi's regime for the treatment of diabetic ulcers (in Chinese) special publicaiton on Diabetic Ulcer. Shanghai Research Institute on TCM.
- [Derived] Leung PC, Pang SY, Wong EL, Cheng KF. Inflammatory state of type II diabetic patients with chronic ulcers in response to herbal treatment. Foot (Edinb). 2012 Sep;22(3):181-5. doi: 10.1016/j.foot.2012.03.001. Epub 2012 Mar 30. PMID 22463944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Apr 2002 to Apr 2006, Orthopaedic Department, Prince of Wales Hospital, HK Apr 2002 to Apr 2006, Orthopaedic Department, Kwong Wah Hospital, HK
Pre-assignment Details: Liver Function and Renal Function test normal. Patients suffering from serious cardiac and renal deficiencies were excluded from the study because of safety measure.
Period: Overall Study
Arm/Group | Traditional Chinese Medicine | Placebo
Started | 40 | 40
Completed | 37 | 31
Not Completed | 3 | 9
Not completed — Physician Decision | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Chinese Medicine | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (12.6) | 68.5 (11.1) | 67.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 25 | 22 | 47
Region of Enrollment [Number; unit: participants]
  Hong Kong | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Limb Salvage
Description: The number of successful limb rescued (without amputation).
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | Traditional Chinese Medicine | Placebo
Number analyzed (Participants) | 40 | 40
Participants | 37 | 31

2. Secondary Outcome: Tumour Necrosis Factor-alpha Levels in Serum
Description: The state of inflammation at baseline and at 4 weeks after treatment. TNF-alpha are in value of serum level.
Time Frame: Baseline and 4 week
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Traditional Chinese Medicine | Placebo
Number analyzed (Participants) | 40 | 40
pg/mL
  Baseline | 48 (116) | 44 (83)
  Week 4 | 28 (62) | 39 (64)

3. Secondary Outcome: Time of Ulcer Healing
Description: Time taken for maturation of granulation to enable skin grafting.
Time Frame: 24 week
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Traditional Chinese Medicine | Placebo
Number analyzed (Participants) | 37 | 31
Weeks | 5.9 (1.4) | 9.2 (1.9)

ADVERSE EVENTS:
Time Frame: 24weeks
Description: During the 24 weeks of treatment, some selflimiting adverse events (epigastric pain, dry month,and diarrhoea) were experienced.
Arm/Group | Traditional Chinese Medicine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No